CLINICAL TRIAL: NCT05149534
Title: Repetitive Transcranial Magnetic Stimulation Augmented Written Exposure Therapy for Veterans With PTSD
Brief Title: rTMS-augmented Written Exposure Therapy for PTSD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: National Center for PTSD (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MHBP-007-20F; 1IK2CX002101-01A2 (NIH)
Record Dates: First submitted 2021-11-24; First posted 2021-12-08 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Post Traumatic Stress Disorder
Keywords: PTSD; Emotion Regulation; Cognitive flexibility; Affective Flexibility; Veterans
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Emotional Regulation | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Double blind, randomized clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants deemed eligible after the baseline assessments will be randomized using a computerized block randomization with a 1:1 allocation ratio of active rTMS/WET and sham rTMS/WET conditions. The investigators will be utilizing permuted block design with randomized blocks of 4 and 2. This will be conducted by an independent study coordinator who will be uninvolved in the research beyond randomization and blinding with assistance from a data analyst in addition to statistics consultant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active TMS/WET (Experimental): Active repetitive transcranial magnetic stimulation completed prior to written exposure therapy
  Interventions: Behavioral: Written Exposure Therapy; Device: repetitive transcranial magnetic stimulation
- Sham TMS/WET (Sham Comparator): Sham repetitive transcranial magnetic stimulation completed prior to written exposure therapy
  Interventions: Behavioral: Written Exposure Therapy; Device: repetitive transcranial magnetic stimulation

INTERVENTIONS:
Behavioral: Written Exposure Therapy — Narrative written disclosure of trauma administered in an evidence-based protocol.
  Other Names: WET
Device: repetitive transcranial magnetic stimulation — Noninvasive magnetic neuromodulation device
  Other Names: rTMS

SUMMARY:
Post-traumatic stress disorder (PTSD) is prevalent and represents a high healthcare burden among Veterans. Repetitive transcranial magnetic stimulation (rTMS) is a brain-based therapy that may be effective for treating PTSD. The theorized mechanism of rTMS is enhancement of emotional flexibility via the dorsolateral prefrontal cortex node of the brain's cognitive control network. Given this mechanism of action, adding rTMS to an evidence-based psychotherapy (EBP) for PTSD may enhance treatment effects. Written exposure therapy (WET) is a brief EBP for PTSD found to reduce attrition compared to lengthier first line treatments. In this study, the investigators will determine if active rTMS added to WET compared with sham rTMS added to WET results in improved PTSD outcomes. The investigators will also determine if emotional flexibility is a mechanism of symptom improvement. This work will improve upon PTSD intervention and inform the mechanism of treatment effectiveness for Veterans suffering from PTSD.

DETAILED DESCRIPTION:
The overarching goal of this CDA-2 proposal is to use repetitive transcranial magnetic stimulation (rTMS) to augment effectiveness of written exposure therapy (WET), a narrative-based trauma exposure paradigm, in treating posttraumatic stress disorder (PTSD) and emotion dysregulation in Operations Enduring Freedom (OEF) and Iraqi Freedom (OIF) Veterans. As a clinical neuropsychologist with expertise in emotion regulation, Dr. Lantrip's long-term goal is to improve upon and develop effective interventions for trauma-related illness in Veterans by identifying and targeting behavioral and neural mechanisms.

OEF/OIF Veterans have experienced increased length and number of deployments, contributing to diagnosis of PTSD. rTMS is a brain-based therapy involving application of a repetitive, brief magnetic pulse to the scalp through an electromagnetic coil. rTMS applied to the dorsolateral prefrontal cortex (DLPFC) has efficacy in patients with treatment-resistant depression, and recent work has shown efficacy for treating PTSD. Standard rTMS treatments are stand-alone, though the unique properties of rTMS may make it more effective when added to a psychotherapy such as an evidence-based psychotherapy (EBP) for PTSD.

rTMS is theorized to act on the DLPFC node of the brain's cognitive control network (CCN) to improve emotion regulatory processes and facilitate reduction in affective symptoms. In support of this theory, studies have found that improvements in affective flexibility, upregulation of positive affect, and downregulation of attention to negative stimuli occur in task-based paradigms immediately following stimulation of the DLPFC with rTMS in a single-session. In addition, recent research has found that rTMS prior to cognitive processing therapy (CPT) in Veterans with PTSD is effective at improving PTSD outcomes compared to sham rTMS plus CPT, possibly through the regulatory mechanism of the CCN. Given these promising findings, further study into optimizing rTMS-augmented EBPs for PTSD is warranted.

There are limitations to both rTMS and first line EBPs for PTSD. One problem is high numbers of sessions needed for effective treatment (i.e. 20 sessions of rTMS and 12-18 sessions of EBPs) contributing to high attrition rates. A large multi-site study of VA patients in PTSD clinic found that just 2% of a sample of 1924 Veterans who had at least one session of EBP received an "adequate dose" of at least 8 sessions.12 A potential optimization for rTMS-augmented EBPs would be to reduce session number to improve retention. WET is a novel EBP for PTSD that is non-inferior to CPT in as few as 5 sessions. Using rTMS to augment WET in Veterans with PTSD is a crucial step in this line of inquiry.

This double-blind, Phase II randomized controlled trial will examine whether rTMS added to WET results in superior outcomes compared to sham rTMS added to WET (N=98 with women and men equally represented). The investigators will randomize 49 OEF/OIF Veterans with PTSD to undergo an active rTMS/WET treatment protocol versus 49 OEF/OIF Veterans given a sham rTMS/WET treatment.

Specific Aim 1: To compare PTSD outcomes of those who experience active rTMS/WET versus sham rTMS/WET. Hypothesis 1: Active rTMS added to WET will contribute to greater PTSD symptom reduction compared to sham rTMS added to WET in Veterans with PTSD.

Specific Aim 2a: If there is a treatment effect in Aim 1, determine if emotional flexibility mediates the rTMS/WET-PTSD relation. Aim 2b (exploratory): Determine if emotional flexibility has a unique mediating effect over cognitive flexibility. Hypothesis 2a: Significant reduction in PTSD symptoms will be partially mediated by emotional flexibility. Hypothesis 2b: Significant reduction in PTSD symptoms will be partially mediated by cognitive flexibility, but to a lesser extent than emotional flexibility.

This CDA-2 extends Dr. Lantrip's research integrating emotion regulation and neurostimulation to understand and improve upon treatment of PTSD in Veterans. The CDA-2 will provide her with specialized training in WET, a unique exposure-based therapy for the treatment of trauma, as well as clinical trials for PTSD, and neurostimulation. The mentoring team integrates expertise in the proposed areas of study and extensive experience mentoring early career investigators. Project findings will inform a future VA Merit proposal, which will focus on individual differences and mechanisms contributing to PTSD symptom improvement in TMS-augmented behavioral therapy. This study has the potential to inform and improve upon existing treatments for PTSD. Together, Dr. Lantrip's work aligns with VA's priorities, CR&D's mission, and with the goal to provide the highest quality of care for Veterans.

ELIGIBILITY:
Inclusion Criteria:

-All veterans are eligible to be included in the study if they meet all the following criteria:

* veteran;
* English-speaking and able to provide written informed consent;
* diagnosed with PTSD;
* between the ages of 18 and 60 years. Participants over age 60 will not be included, as aging is known to impact brain structure, and thus the potential accuracy of the rTMS target, independently of PTSD.

Exclusion Criteria:

* Individuals with history of seizures or other serious neurological history including acquired, developmental or degenerative neurologic illness, identified through medical chart review, will be excluded due to potential lowered threshold for seizures during rTMS stimulation.
* The effects of rTMS are unknown on fetal development, therefore, women who are pregnant will be excluded.
* Participants will also be screened and excluded if any of the following are met:

  * current psychosis including psychotic disorder,
  * bipolar disorder,
  * schizophrenia; or another severe cognitive or psychiatric disorder;
  * positive screen for current suicidal intent and plan [with a score of 2 or 3 on BDI-2 item 9];
  * current substance use disorder; or substance use in the last 12 hours before the rTMS session.
* The investigators note that PTSD is often comorbid with traumatic brain injury (TBI) in military veterans who were deployed to a war zone. The investigators will use the Department of Defense and Veterans Affairs consensus-based classification of TBI severity for classification of TBI.
* Participants with moderate or severe TBI will be excluded.
* Participants with mild traumatic brain injury (mTBI) or concussion will be enrolled. This will enhance the ecological validity of the study.
* Participants with cognitive impairment as evidenced by a Montreal Cognitive Screen (MoCA) less than 23/30 or estimated baseline intellectual ability of a standard score of less than 80 on a word reading test will be excluded due to potential neurocognitive differences.
* Participants on psychotropic medications will not be excluded, but participants will be required to be stable on their medication for at least four weeks prior to beginning the study and throughout the time of study.
* Participants enrolled in long term, supportive psychotherapy (i.e. not an evidence-based psychotherapy (EBP)) may continue to be involved in their treatment throughout the study. However, participants involved in a concurrent EBPs will be excluded. Participants will be asked to disclose whether they chose to participate in an EBP during the course of the treatment or followup phases of the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 98 (Estimated)
Dates: Start 2022-01-03 (Actual); Primary Completion 2027-01-29 (Estimated); Study Completion 2027-01-29 (Estimated)

PRIMARY OUTCOMES:
Change in Clinician Administered PTSD Scale for DSM-5 (CAPS-5) | Pre intervention (Baseline), post-intervention (Treatment Session 5), and following the conclusion of the intervention, up to 3 months
  The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) is a 30-item structured interview designed to make both a current and lifetime diagnosis of PTSD and to assess PTSD symptom severity over the last week or month. The assessor combines information about frequency and intensity of an item into a single severity rating. CAPS-5 total symptom severity scores are calculated by summing the individual item scores for symptoms corresponding to a given DSM-5 cluster. Severity ratings are from 0 (absent) to 5 (extreme/incapacitating)

SECONDARY OUTCOMES:
Change in PTSD Symptom Checklist for DSM-5 (PCL-5) | Pre intervention (Baseline), post-intervention (Treatment Session 5), and following the conclusion of the intervention, up to 3 months
  PTSD will be measured with the widely used 20-item Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5), which assesses severity of each DSM-5 PTSD symptom using a Likert-style ranging from 0 (not at all) to 4 (extreme). A total score of 31-33 is suggestive of a PTSD diagnosis. Change in PTSD symptom severity from pre-to post-intervention will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Crystal M Lantrip, Principal Investigator — Central Texas Veterans Health Care System, Temple, TX
Locations (1):
- Central Texas Veterans Health Care System, Temple, TX, Temple, Texas, United States

IPD SHARING:
Plan to Share IPD: No
A Limited Dataset (LDS) will be created and shared pursuant to a Data Use Agreement (DUA) appropriately limiting use of the dataset and prohibiting the recipient from identifying or re-identifying (or taking steps to identify or re-identify) any individual whose data are included in the dataset.